CLINICAL TRIAL: NCT00361205
Title: Electronic Compliance Monitoring in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Collaborators: Neurosciences Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003/03
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2005-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease, pharmacology, compliance, dopaminergic
MeSH Terms: conditions — Parkinson Disease; Patient Compliance

INTERVENTIONS:
Device: Electronic Monitoring cap

SUMMARY:
Patients with Parkinson's Disease (PD) depend on medication for relief of motor symptoms, and for this reason are often assumed to medicate very carefully. Overall, medication adherence is very good, but a subset of 15 to 20% of cases take less than 80% of the total prescribed dose. However, irregular timing of drug ingestion is almost universal, perhaps contributed by fluctuating symptoms and drug regimen complexity. Pulsatile dopaminergic stimulation in the basal ganglia is implicated in the development and manifestation of motor complications of advancing PD. Irregular medication intake is likely to contribute to peaks and troughs in serum and brain drug levels. In other diseases, patient adherence to prescribed medication improves through simplifying drug regimens, providing additional education, counselling and behavioural approaches and providing reminder packaging. We tested the effect on the timing of medicine ingestion of an educational approach, in which patients were given detailed additional information about the continuous dopaminergic theory.

DETAILED DESCRIPTION:
Patients attending a regional movement disorder clinic with idiopathic PD (by UK Brain Bank criteria) and prescribed one or more antiparkinson drug (including dopamine agonist or levodopa) were invited to participate. Patients who were unable to manipulate the electronic pill monitoring bottles, or whose compliance would be adversely affected by using the electronic pill monitoring bottles (e.g. those reliant on a compliance aid) were excluded. The study received ethics approval and signed consent was obtained. During the study medication was adjusted according to clinical need. The increase in levodopa equivalent units during the study period was calculated according to established formula[12].

Baseline assessments of unified Parkinson's disease rating scale (UPDRS), Hoehn and Yahr, Schwab and England, mini-mental state examination, geriatric depression scale and quality of life score (PDQ 39) were performed. Clinical scoring was blind to patient group and performed in an 'on' state. The UPDRS 3 and adverse events were recorded at each visit. The quality of life score (PDQ 39) was repeated at the final visit.

All antiparkinson drugs were monitored during two 3 month periods (before and after the educational intervention) using electronic monitoring pill bottles (MEMS®, Aardex, Switzerland), a device which records the time and date of bottle opening.

Patients randomly assigned (computer generated and placed in opaque envelopes) to the active (counselled) group were given verbal and written information about the continuous dopaminergic theory, and written advice on optimal medicine timing tailored to their own drug regimen. The counselling explained that in health, brain dopamine is constant, and that fluctuations from Parkinson's medications should be minimised to simulate normal dopamine levels. Control patients received standard care, but also had medication intake monitored using the MEMS device.

Timing compliance (the percentage of doses taken at the correct time interval) was calculated using time intervals which optimise the pharmacokinetic profile, plus a 25% allowance, eg. 3 times daily medication is satisfactory at between 6 and 10 hours. Selegiline 5mg twice daily was excluded from analysis as the second dose is taken at lunchtime to avoid sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women between 18 and 80 years.
* Patient has idiopathic Parkinson's Disease according to Brain Bank criteria. Reference Hughes A J, Daniel S E, Kilford L, Lees A J, Accuracy of Clinical Diagnosis of Idiopathic Parkinson's disease; A clinical Pathological study of 100 cases, JNNP 1992, 55(3): 181 - 184
* Patient is on stable doses of anti-Parkinson's disease medication, which are not expected to change during the study period.
* Patient is taking levodopa and/or dopamine agonist treatment.
* Patient (assisted by a carer where appropriate) is able to take their medication using the MEMS (electronic monitoring) containers.
* Patients using a dosette box or similar device for their medication are willing to use the MEMS containers for their PD medication
* The investigator judges that the patient's care and symptom control will not be adversely affected by entering the study and using the MEMS device.

Exclusion Criteria:

* Patient is taking anti-Parkinson's disease therapy intermittently or on "as required" basis (such as rescue therapy for off periods). Intermittent Domperidone is allowed.
* Severe co-morbid condition such as severe heart, liver, or kidney disease or cancer diagnosis where the co-morbid condition is of greater health significance than the Parkinson's disease in terms of life expectancy and levels of care required.
* Patient is expected to undergo hospital admission during the study period (such as elective surgery).
* Patient is on non standard drug treatment / combination therapy. This would include e.g. a combination of 2 different oral dopamine agonists, doses of dopamine agonist taken at higher than recommended for routine practice.
* New antiparkinson treatment is being introduced at the time of recruitment or during the one month monitoring period.
* Patient is taking only adjunct therapy (eg. Selegiline, Amantadine, anticholinergic therapy).
* Patient is taking part in a clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-11; Study Completion 2005-09

PRIMARY OUTCOMES:
Timing compliance

SECONDARY OUTCOMES:
Parkinson motor scores

CONTACTS AND LOCATIONS:
Overall Officials: Donald Grosset, MBChB, MD, Principal Investigator

REFERENCES:
- [Derived] Grosset KA, Grosset DG. Effect of educational intervention on medication timing in Parkinson's disease: a randomized controlled trial. BMC Neurol. 2007 Jul 16;7:20. doi: 10.1186/1471-2377-7-20. PMID 17634109